CLINICAL TRIAL: NCT06756828
Title: Study on Regional Structural Changes in the Cerebellum Associated with Blood Biomarkers, Cognitive Decline, and Physical Performance in Alzheimer's Spectrum Patients Following a 3-Month Melatonin Treatment Using Digital Health Technology
Brief Title: Effects of 3-Month Melatonin Treatment on Regional Cerebellar Structure and Blood Biomarkers in Alzheimer's Disease Spectrum
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VC24OISI0285
Record Dates: First submitted 2024-12-03; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Elderly; Alzheimer Disease; Melatonin; Cognitive Decline; Biomarker with Neurodegeneration Patients; Cerebellum
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin group (Experimental): Taking 2mg of melatonin 2 hours before going to bed for 12 weeks.
  Interventions: Drug: Melatonin
- Cognitive behavioral therapy group (Other): 15minutes of sleep hygiene education on the first day of visiting the hospital
  Interventions: Behavioral: Cognitive behavioral therapy group for insomnia

INTERVENTIONS:
Drug: Melatonin — 3months melatonin
  Arms: Melatonin group
Behavioral: Cognitive behavioral therapy group for insomnia — 15minutes of sleep hygiene education on the first day of visiting the hospital
  Arms: Cognitive behavioral therapy group

SUMMARY:
The goal of this clinical trial is to explore and verify the preventive effects of melatonin on the progression of Alzheimer's disease. The study aims to analyze the changes in blood biomarkers (phosphorylated tau, glial fibrillary acidic protein, neurofilament chain), various sleep-related subjective report questionnaire scores, physical performance, cognitive function scores and cerebellar volume change after three months of melatonin administration in patients with Alzheimer's-type mild cognitive impairment (MCI) accompanied by insomnia. The main questions it aims to answer are:

1. Does melatonin administration alter the levels of blood biomarkers associated with Alzheimer's disease?
2. What changes occur in sleep-related subjective report questionnaire scores and cognitive function scores following melatonin administration?
3. Does melatonin administration effect on physical performance?
4. Is there any relations between cognitive decline, phsycal performance and cerebellar volume change? We will compare the data collected before and after melatonin administration to determine its preventive effects on Alzheimer's disease progression.

Participants Will:

1. Take melatonin every day for 3 months and Complete sleep-related subjective report questionnaires, neuropsychological assessments and physical performance test
2. Visit the clinic at the initial visit and after 3 months for checkups and tests.
3. Complete sleep-related subjective report questionnaires and neuropsychological assessments and physical performance test
4. Provide blood samples for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 60 to 90 years
* Individuals presenting with cognitive impairment as their chief complaint at the Department of Psychiatry, St. Vincent's Hospital
* Those capable of undergoing imaging studies, including Brain MRI and Amyloid PET CT
* Individuals able to complete cognitive function tests, such as the Alzheimer's Disease Consortium test battery, K-MMSE, CDR, and GDS
* Participants who can perform tests at the hospital's Smart Center, including the Short Physical Performance Battery and body composition analysis using direct segmental multi-frequency bioelectrical impedance analysis for sarcopenia
* Individuals on acetylcholinesterase inhibitors (ACEi) or NMDA receptor antagonists who have maintained the same dosage and regimen for more than 3 months from the screening date.
* Patients who are taking medications for cognitive function treatment other than acetylcholinesterase inhibitors and NMDA receptor antagonists (e.g., pregabalin, gabapentin, choline alfoscerate), as well as medications for chronic diseases such as antidepressants, antihypertensives, diabetes, hyperlipidemia, thyroid disorders, etc., must have maintained the same dosage and regimen for more than 1 month from the screening date.
* Individuals with sufficient language proficiency to read and understand the informed consent document and respond to survey questionnaires

Exclusion Criteria:

* Individuals with progressive mental or neurological disorders (including those with a history of psychotic disorders such as major depressive disorder, bipolar disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, or unspecified psychosis; patients currently experiencing major depressive disorder with psychotic symptoms; organic mental disorders; epilepsy or seizure disorders; patients currently suffering from eating disorders or obsessive-compulsive disorder).
* Individuals with unstable or severe medical conditions.
* Patients with severe snoring, REM sleep behavior disorder, or narcolepsy.
* Illiterate individuals.
* Individuals who, in the opinion of the investigator, are deemed unable to comply with the requirements of the study.
* Patients currently taking sleeping pills within 2 weeks of the screening point.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum p-Tau 217 Levels from Baseline to Week 12 | Baseline and Week 12
  Serum p-Tau 217 levels will be measured at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in concentration (pg/mL) between baseline and Week 12.
Change in Serum Glial Fibrillary Acidic Protein (GFAP) Levels from Baseline to Week 12 | Baseline and Week 12
  Serum GFAP levels will be measured at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in concentration (pg/mL) between baseline and Week 12
Change in Serum Neurofilament Light Chain (NfL) Levels from Baseline to Week 12 | Baseline and Week 12
  Serum Neurofilament Light Chain (NfL) levels will be measured at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in concentration (pg/mL) between baseline and Week 12.
Change in Physical Performance from Baseline to Week 12 | Baseline and Week 12
  Physical performance will be assessed using the Short Physical Performance Battery (SPPB), which evaluates balance, gait speed, and lower body strength. Changes will be reported as differences in total SPPB scores(points) between baseline and Week 12.

SECONDARY OUTCOMES:
Change in Global Deterioration Scale (GDS) Scores from Baseline to Week 12 | Baseline and Week 12
  Global Deterioration Scale (GDS) scores will be assessed as a measure of cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Clinical Dementia Rating (CDR) Scores from Baseline to Week 12 | Baseline and Week 12
  Clinical Dementia Rating (CDR) scores will be assessed as a measure of cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Verbal Fluency Scores from Baseline to Week 12 | Baseline and Week 12
  Verbal fluency(points), assessed as a subtest of the CERAD-K battery, will be used to measure cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Mini-Mental State Examination (MMSE) Scores from Baseline to Week 12 | Baseline and Week 12
  The Mini-Mental State Examination (MMSE)(points), assessed as a subtest of the CERAD-K battery, will be used to measure cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Boston Naming Test (BNT) Scores from Baseline to Week 12 | Baseline and Week 12
  The Boston Naming Test (BNT)(points), assessed as a subtest of the CERAD-K battery, will be used to evaluate cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Word List Recall Scores from Baseline to Week 12 | Baseline and Week 12
  Word List Recall(points), assessed as a subtest of the CERAD-K battery, will be used to evaluate cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Word List Recognition Scores from Baseline to Week 12 | Baseline and Week 12
  Word List Recognition(points), assessed as a subtest of the CERAD-K battery, will be used to evaluate cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Constructional recall from Baseline to Week 12 | Baseline and Week 12
  Constructional recall(points), assessed as a subtest of the CERAD-K battery, will be used to evaluate cognitive function at baseline and at the end of the 12-week treatment period. Changes will be reported as the difference in scores between baseline and Week 12.
Change in Pittsburgh Sleep Quality Index (PSQI) Global Scores from Baseline to Week 12 | Baseline and Week 12
  The Pittsburgh Sleep Quality Index (PSQI) global score will be used to assess sleep quality. A global score greater than 5 indicates significant sleep disturbances, with higher scores representing greater levels of sleep disturbance. Changes will be reported as the difference in PSQI global scores between baseline and Week 12.
Change in Insomnia Severity Index (ISI) Scores from Baseline to Week 12 | Baseline and Week 12
  The Insomnia Severity Index (ISI) is a brief, self-rated scale consisting of seven items scored on a 0-4 scale, used to measure the severity of insomnia.Scores of 15 or higher indicate moderate to severe insomnia. Changes will be reported as the difference in ISI scores between baseline and Week 12.
Change in Epworth Sleepiness Scale (ESS) Scores from Baseline to Week 12 | Baseline and Week 12
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire consisting of eight items designed to measure daytime sleepiness in daily life. Scores above 10 indicate clinically meaningful daytime sleepiness, with higher scores reflecting greater severity. Changes will be reported as the difference in ESS scores between baseline and Week 12.
Differences in Cerebellum Volume and Its Correlation with Blood Biomarkers, Physical Performance, Cognitive Tests, and Sleep Questionnaire Responses | At the time of enrollment
  The study will assess cerebellum volume at the time of enrollment and analyze its correlations with blood biomarker levels (p-Tau 217, NfL), physical performance metrics, cognitive test scores, and sleep-related questionnaire responses. Correlations will be reported using Spearman's correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Yoo Hyun Um Um, Assitant professor, Ph.D, MD, Principal Investigator — St.Vincent's Hospital, College of Medicine, Catholic University of Korea